CLINICAL TRIAL: NCT06502899
Title: Prognostic Value of CMR-related Parameters in Patients with MINOCA
Brief Title: CMR in Myocardial Infarction with Nonobstructive Coronary Arteries
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CMR in MINOCA
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Magnetic Resonance; Myocardial Infarction with Nonobstructive Coronary Arteries; Strain; Extracellular Volume
MeSH Terms: conditions — MINOCA; Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- diagnosed with MINOCA and completed with cardiac magnetic resonance
  Interventions: Other: Cardiac MRI

INTERVENTIONS:
Other: Cardiac MRI — Patients with a diagnosis of MINOCA and completed CMR were included in this study

SUMMARY:
MINOCA is accompanied by a worse prognosis, which is related to the inability to clarify the etiology.CMR has been explicitly recommended by guidelines as an etiologic diagnostic tool for MINOCA. Although CMR-related parameters, such as strain and ECV, have been shown to be associated with prognosis in patients with myocardial infarction. However, the relationship between CMR-strain or ECV and MINOCA is unclear. The aim of this study was to investigate the characterization of CMR-strain or ECV in patients with MINOCA and the relationship with prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Complete CMR during hospitalization;
2. CAG results suggesting coronary stenosis of less than 50%;
3. peak hsTnT above the 99th percentile.

Exclusion Criteria:

* CMR image sequences are missing or of poor quality.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We consecutively selected patients who were suspected of myocardial infarction with concomitant CAG from January 2019 to June 2024 at the Affiliated Hospital of Xuzhou Medical University. All patients completed CMR during hospitalization. hsTnT peak was above the 99th percentile and CAG less than 50% in all patients.
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Primary endpoint events included any cause, non-fatal infarction, stroke, or cardiac readmission. | All patients were followed until June 30, 2024

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Considering the patient's privacy and the next steps in our research program

REFERENCES:
- [Derived] Abdu FA, Chen L, Qiu B, Liu L, Mohammed AQ, Lv X, Yin G, Zhang W, Alifu J, Chen W, Lu Y, Che W. Prognostic Impact of Infarct Size and Coronary Microvascular Function Via Cardiovascular Magnetic Resonance and Coronary Angiography-Derived Index of Microcirculatory Resistance in Myocardial Infarction With Nonobstructive Coronary Arteries. J Am Heart Assoc. 2026 Jan 6;15(1):e043169. doi: 10.1161/JAHA.125.043169. Epub 2025 Dec 18. PMID 41413401
- [Derived] Chen L, Ge L, Abdu FA, Du X, Liu J, Chen W, Lu Y, Che W. Prognostic value of CMR-derived extracellular volume in myocardial infarction with non-obstructive coronary arteries. Int J Cardiol. 2025 Oct 15;437:133528. doi: 10.1016/j.ijcard.2025.133528. Epub 2025 Jun 18. PMID 40541789
- [Derived] Chen L, Qiu B, Abdu FA, Liu L, Zhang W, Wang C, Alifu J, Qi P, Che W, Lu Y. Prognostic Value of Strain by Tissue Tracking Cardiac Magnetic Resonance in Myocardial Infarction With Nonobstructive Coronary Arteries. J Am Heart Assoc. 2025 Apr 15;14(8):e039395. doi: 10.1161/JAHA.124.039395. Epub 2025 Apr 7. PMID 40194976